CLINICAL TRIAL: NCT00401271
Title: A Phase II Trial to Evaluate the Safety, Efficacy and Pharmacokinetics of Four Oral Doses of OPC-67683 in Patients With Uncomplicated, Smear-Positive, Pulmonary Tuberculosis
Brief Title: Safety, Efficacy and Pharmacokinetics of OPC-67683 in Patients With Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Frankfurt Research Institute GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 242-06-101
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2007-03-07 (Estimated); Status verified 2007-03

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — OPC-67683

INTERVENTIONS:
Drug: OPC-67683
Drug: Rifafour e-275

SUMMARY:
The purpose of this trial is to evaluate the safety, efficacy and pharmacokinetics of 100mg, 200mg , 300mg and 400mg once daily of OPC-67683, administered orally for 14 consecutive days, in patients with uncomplicated, smear-positive pulmonary TB.

The four OPC-67683 treatment groups will comprise 12 patients each and the one standard therapy (Rifafour e-275) group six patients.

Trial 242-06-101 is an exploratory and not a confirmatory trial and as such no hypothesis will be tested statistically.

The control group, six patients treated with Rifafour, will serve as an control to confirm the microbiological assessments during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all trial-related procedures.
* Male and female patients aged between 18 and 64 years, inclusive.
* Newly diagnosed, previously untreated, uncomplicated, smear positive, pulmonary TB.
* A chest X-ray finding compatible with TB.
* Sputum positive on direct microscopy for acid-fast bacilli (AFB) (at least 1+).
* Able to produce an adequate volume of sputum (10mL or more estimated overnight production).
* Female patients of childbearing potential must demonstrate a negative pregnancy test result. Furthermore they must agree to use a highly effective method of contraception.
* Male patients must agree to use an adequate method of contraception.

Exclusion Criteria:

* Poor general condition where no delay in treatment can be tolerated or where immediate hospital admission is warranted.
* Rifampicin-resistant bacteria detected in the sputum susceptibility testing at Screening.
* Treatment received with any drug active against M. tuberculosis within the 3 months prior to Screening.
* History of allergy to any nitro-imidazole derivates, rifamycin derivatives, isoniazid derivatives, pyrazinamide or ethambutol.
* Clinical evidence of severe extrathoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis).
* Evidence of pulmonary silicosis, lung fibrosis, or other lung condition considered as severe by the investigator (other than TB).
* Presence of chronic obstructive pulmonary disease or asthma.
* Any clinically relevant concomitant conditions or renal impairment characterized by serum creatinine levels >= 1.5xULN or hepatic impairment or alcohol abuse characterized by ALT and/or aspartate transferase (AST) levels 3xULN and/or gamma-glutamyl transpeptidase (GGT) levels 3xULN of the laboratory reference range.
* Known or suspected alcohol or drug abuse, that is, abuse sufficient enough to compromise the safety or cooperation of the patient, in the opinion of the investigator, and as evident by a positive urine drug screen.
* Neuropathy, psychosis or epilepsy.
* Clinically relevant changes in the ECG such as atrioventricular (AV) block, prolongation of the QRS complex >120 milliseconds (in both male and female patients), or QTcB interval >430 milliseconds in male patients and >450 milliseconds in female patients. Family history of long QT syndromes and/or Torsade de Pointes.
* History of or current clinically relevant cardiovascular disorder such as hypokalaemia, heart failure, coronary heart disease, hypertension, arrhythmia or symptom strongly suggestive of such a problem (for example, syncope or palpitations), tachyarrhythmia or status after myocardial infarction.
* Known bleeding disorders or family history of bleeding disorders.
* Diabetes treated with insulin.
* Evidence of clinically significant metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied).
* Any diseases or conditions in which the use of rifampicin, isoniazid, pyrazinamide or ethambutol is contra-indicated.
* Any disease or conditions in which any of the medicinal products listed in the protocol, is used. Treatment received with quinolones and prednisolone within 3 months prior to Screening.
* Administration of an IMP within 1 month prior to Screening.
* Pregnancy, breast-feeding, or planning to conceive or father a child within the timeframe described in the informed consent form.
* Recent use of methadone, benzodiazepines, cocaine, amphetamine/metamphetamine, tetrahydrocannabinol, barbiturates, tricyclic antidepressants, and opiates as determined by a urine drug screen.
* Helper/inducer T lymphocyte (CD4 cell) count of <=350x106/L.
* Use of antiretroviral therapy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54
Dates: Start 2006-11; Study Completion 2007-03

PRIMARY OUTCOMES:
TB bacterial load in sputum measured as colony forming units

SECONDARY OUTCOMES:
Early Bactericidal Activity (EBA)
Slope 0-14
Tme to culture positivity

CONTACTS AND LOCATIONS:
Overall Officials: Andreas H Diacon, Dr., Principal Investigator — Tiervlei Trial Center; Roxana Rustomjee, Dr., Principal Investigator — Medical Research Council; Rodney Dawson, Dr., Principal Investigator — University of Cape Town Lung Institute
Locations (3):
- South Africa (3):
  - Tiervlei Trial Center, Karl Bremer Hospital, Bellville, W Cape
  - University of Cape Town Lung Institute, Mowbray, W Cape
  - Medical Research Council, Durban